CLINICAL TRIAL: NCT00224367
Title: Does Early Ambulation After Hip Fracture Surgery Accelerate Recovery?: A Randomised Controlled Trial
Brief Title: Does Early Ambulation After Hip Fracture Surgery Accelerate Recovery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: T10414; Award number A33429
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2005-09-23 (Estimated); Status verified 2005-02

CONDITIONS: Fractured Hip
Keywords: fracture; hip; ambulation
MeSH Terms: conditions — Hip Fractures; Fractures, Bone

INTERVENTIONS:
Behavioral: time to first ambulation

SUMMARY:
Hip fractures are a significant problem for healthcare providers due to the increasing incidence of fractures in an ageing population. Hip fracture is the most frequent fracture for people over 80 years of age and the second most frequent for those over 65 years. It is projected that by 2051, 23% of the Australian population will be older than 65 and the number of hip fractures will rise fourfold (17,000 in 2004, to 60,000 in 2051).

Evidence-based clinical practice guidelines regarding management of hip fracture were published in the Medical Journal of Australia in 1999 and updated in 2003. Seventeen aspects of treatment were systematically reviewed, including mobilisation after surgery. Early assisted ambulation within 48 hours post surgery was recommended (Chilov 2003 p 490). However, the recommendation was based on observational (level 3) evidence only.

Early mobilization post surgery is resource intensive. Early mobilization is challenging and uncomfortable for the patient and requires the assistance of one or sometimes two, physiotherapists available seven days per week. Benefits must be rigorously evaluated to justify recommendation. We undertook a randomized controlled trial of the effect of two different 'time to first ambulation' intervals after hip fracture surgery on patient and hospital outcomes.Our hypothesis was that early mobilisation would accelerate functional recovery after hip fracture surgery.

DETAILED DESCRIPTION:
Methods Inclusions: Consecutive patients admitted via the emergency department to The Alfred hospital Melbourne, for surgical fixation of an acute fracture of the hip (by a compression screw and plate or a hemiarthroplasty).

Exclusions:fracture was pathological, postoperative orders were for non-weight bearing on the operated hip, the patient was admitted from a nursing home or the patient was non-ambulant pre-morbidly.

Sixty eligible patients were randomly allocated, using a computer generated program, into one of two groups.

Management All patients received routine, standard post-operative medical and nursing clinical care, as currently practiced at The Alfred. All patients were transferred to sit out of bed as early as possible after surgery.

Ambulation The physiotherapy ambulation re-education program was implemented once per day over 7 days for all participants. The time to first walk differed between the groups.

Data collection On admission: gender, age, preoperative mobility, social supports, mental ability and medical comorbidity,pre-existing medical comorbidity (cardiac, respiratory, neurological, diabetes) and mental ability.

Additional data from each patients medical record including: type of surgical fixation (nail/screw and plate, hemi-arthroplasty), wait time to surgery, time surgery completed, and time to first sit out of bed and time to first walk.

Outcome measures The primary outcome measure was the patient's functional level, represented by the distance they walked and the level of assistance required to transfer from supine to sit and sit to stand and to negotiate one step, on day-7 post surgery.

Secondary outcome measures included discharge destination and length of stay in the acute care (days from admission to discharge from The Alfred).

Data analysis Statistical analysis was performed using SAS version 8.2. (SAS Institute Inc.,Carv, NC, USA). Continuous variables were compared using student t-tests and validated using Wilcoxon rank sum tests. Categorical variables were compared using chi-square tests for equal proportion. A two-sided p-value of 0.05 was considered to be statistically significant.

Sample size A difference between groups equivalent to one standard deviation was perceived to be of clinical importance. With 30 subjects per group, this study had a 97% power to detect a difference equal to one standard deviation with a two-sided p-value of 0.05. A minimum of 16 subjects per subgroup was required for this study to have an 80% power to detect a difference equal to one standard deviation with a two-sided p-value of 0.05.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients admitted via the emergency department to The Alfred hospital Melbourne, for surgical fixation of an acute fracture of the hip (by a compression screw and plate or a hemiarthroplasty) -

Exclusion Criteria:

fracture was pathological, postoperative orders were for non-weight bearing on the operated hip, the patient was admitted from a nursing home or the patient was non-ambulant pre-morbidly. -

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2004-02; Study Completion 2004-12

PRIMARY OUTCOMES:
functional outcome day 7 post-operation

SECONDARY OUTCOMES:
discharge destination
length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Leonie B Oldmeadow, D.Physio, Principal Investigator — The Alfred
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134